CLINICAL TRIAL: NCT03020069
Title: Use of Continuous Glucose Monitoring System With Intensive Feedback in Adolescents With Poorly Controlled Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-01011
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Adolescents; Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Glucose Meter (Experimental): Continuing Glucose Monitoring Device
  Interventions: Device: CGMS Device
- No Glucose Meter (Active Comparator): Average Blood glucose measure
  Interventions: Other: No Device

INTERVENTIONS:
Device: CGMS Device
  Other Names: Continuing Glucose Monitoring Device
  Arms: Glucose Meter
Other: No Device
  Arms: No Glucose Meter

SUMMARY:
The purpose of this study is to determine that continuous glucose monitoring systems (CGMS) with intensive real time feedback about diabetes management from medical staff to the patient will affect motivation and/or behavior, in adolescents with poorly controlled type 1 diabetes. The investigators hypothesize that short-term CGMS use with feedback (and/or lack thereof) and patients' sense of self-efficacy will influence their stage of change and potentially glucose levels.

DETAILED DESCRIPTION:
Sixty adolescents, ages 13-19 years, with type 1 diabetes and an HbA1c > = 8 % who are also naive to CGMS use will be recruited from the diabetes outpatient population followed at Bellevue Hospital, Lutheran Hospital, Woodhull Hospital, and the NYU Fink Pediatric Ambulatory Care Center. Forty subjects will be randomly assigned to the CGMS group and 20 subjects will be assigned to the control group.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes
* HbA1c > = 8 %
* naive to CGMS use

Exclusion Criteria:

* Patients with developmental delay
* Patients who do not use a glucose meter to test capillary blood glucose level
* Patients without access to a telephone will be excluded.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonita Franklin, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- New York University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Glucose Meter: Continuing Glucose Monitoring Device
  CGMS Device
- No Glucose Meter: Average Blood glucose measure
  No Device
Period: Overall Study
Arm/Group | Glucose Meter | No Glucose Meter
Started | 9 | 4
Completed | 9 | 3
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glucose Meter | No Glucose Meter | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Continuous [Median (Full Range); unit: years] | 16 [14 to 18] | 17 [16 to 18] | 16 [14 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Score of Pediatric Quality of Life Inventory 3.2 Diabetes Module (Peds QL 3.2) From Baseline to 3 Months
Description: The PedsQL 3.2 Diabetes Module is composed of 33 items. Item scaling is a 5-point scale from 0 (never) to 4 (almost always). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. The total score is calculated as the sum of all items over the number of items answered on all the scales (total score ranges from 0-3300). Higher scores indicate lower problems. The change in total score is calculated by subtracting the total score at baseline from the total score at 3 months.
Time Frame: Baseline, 3 Months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Glucose Meter | No Glucose Meter
Number analyzed (Participants) | 9 | 3
score on a scale | 6.4 [-11.4 to 15.9] | -3.8 [-21.2 to 4.5]

2. Primary Outcome: Change in Glycated Hemoglobin (HbA1c) Levels From Baseline to 3 Months
Description: HbA1c measurements will be measured in the lab at the location of the patient's visit at baseline and 3 months. The measured HbA1c level at 3 months will be subtracted from the measured level at baseline to calculate the change.
Time Frame: Baseline, 3 Months
Measure: Mean (Full Range); unit: mmol/mol
Arm/Group | Glucose Meter | No Glucose Meter
Number analyzed (Participants) | 9 | 3
mmol/mol | -9.4 [-132 to 67] | -36 [-194 to 24]

3. Primary Outcome: Change in Level of Blood Sugar (Glucose) From Baseline to 3 Months
Description: Blood sugar (glucose) will be measured via glucose monitors. The change in level of blood sugar will be calculated by subtracting the blood glucose level at 3 months from the blood glucose level at baseline.
Time Frame: Baseline, 3 Months
Measure: Mean (Full Range); unit: mg/dl
Arm/Group | Glucose Meter | No Glucose Meter
Number analyzed (Participants) | 9 | 3
mg/dl | -0.1 [-18.3 to 0.7] | 0 [-0.1 to 0.3]

4. Primary Outcome: Change in Score of Diabetes Empowerment Scale Short Form (DES-SF) From Baseline to 3 Months
Description: There are 8 items that constitute the DES-SF. The scale is scored by averaging the scores of all completed items. 1 = strongly disagree and 5 = strongly agree. The change in score between baseline and 3 months will be calculated by subtracting the average score from 3 months from the baseline score.
Time Frame: Baseline, 3 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Glucose Meter | No Glucose Meter
Number analyzed (Participants) | 9 | 3
units on a scale | 0.375 [-.375 to 0.875] | -0.25 [-0.625 to 0]

ADVERSE EVENTS:
Time Frame: For 3 months after randomization
Arm/Group | Glucose Meter | No Glucose Meter
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 0/9 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT03020069/Prot_SAP_000.pdf